CLINICAL TRIAL: NCT02469870
Title: ASD Parent Trainer: Online Coaching for Parents of Children With Autism
Acronym: APT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRIS Media Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2R44MH102845-02 (NIH)
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Autism Disorder
Keywords: Parents of children who have autism; video-conferencing; Applied Behavior Analysis; Acceptance Commitment Training; optimism training; Positive Behavior Support
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autism Parent Trainer (APT) (Experimental): Practiced Routines was a facilitated program. It was organized into four modules that included a total of seven videos ranging from 3-13 minutes each. The topics overlapped with those in the TR program, but included more explicit information on function-based strategies, as well as mindfulness practice. Participants were assigned six fillable forms, and provided supplemental data collection tools. Additional resources focused on mindfulness and PBS within family routines. Eighteen brief guided audio meditations were available to participants via the Practiced MindTM mobile application. The meditations focused on bringing the parents' awareness to both internal and external experiences and helping them act intentionally.
  Interventions: Behavioral: Autism Parent Trainer (APT)
- Teaching Routines (Control (Active Comparator): Teaching Routines was entirely self-directed. The program included eight modules with videos for each ranging 3 - 5 minutes in duration. The topics were antecedent-behavior-consequence method, creating task analyses, antecedent-based strategies, communication, reinforcement, teaching methods, and overcoming obstacles. Participants were assigned six activities using fillable forms and provided additional resources including examples, a glossary of terms, and a list of websites. No feedback was given to the parents apart from the automated completion responses. The participants were given access to the TR LMS for the duration of the study, but post and follow-up assessments were completed at 6 and 10 weeks (i.e., same as the PR condition).
  Interventions: Behavioral: Teaching Routines (Control)

INTERVENTIONS:
Behavioral: Autism Parent Trainer (APT) — Experimental condition
  Arms: Autism Parent Trainer (APT)
Behavioral: Teaching Routines (Control) — Content comparison group.
  Arms: Teaching Routines (Control

SUMMARY:
The evaluation of the program efficacy will be conducted via a randomized control study with 136 parents of children aged 3-8 who have autism. Investigators will test whether, compared to a content comparison group (CC), administration of the APT program over a 3-week intervention period (a) improves child behaviors, (b) increases perceived quality of life, (c) decreases parental stress, (d) increases positive parenting practices, and (e) increases parent knowledge of evidence-based support practices.

DETAILED DESCRIPTION:
Participants. The sample will consist of parents who have at least one child diagnosed with autism (aged 3 to 8) and have access to the Internet. From investigators experience in the Phase I and similar studies, an attrition rate of less than 30% is expected. 180 parents (90 per condition) will ensure that the final sample will be no fewer than 136, with 68 in each condition. Participation will be open to two-parent and single-parent families; only one parent per family will be invited to participate in data collection. No parental age, gender, or race exclusions will apply.

Procedure. All research will be conducted online. IRIS Ed has extensive experience conducting online studies, and has developed successful recruitment, retention, and assessment procedures. Screening, consent, and data collection will be conducted using Qualtrics (see Human Subjects). Google+ Hangouts will be used to conduct the interactive APT training. The CC training materials will be hosted on irisEd.com. Additional training materials will be hosted on YouTube and SoundCloud. Participants will be recruited nationally using approaches and resources that have yielded results in past online interventions.

The APT study will adhere to the following procedures: potential participants will be directed to the recruitment website on Qualtrics and will be screened for eligibility on the following inclusion criteria: (a) have a child aged 3-8 diagnosed with autism and living with the parent, (b) have access to email and an Internet connection, and (c) have access to a computer or other mobile device with a camera and a microphone. Eligible participants will be given a brief explanation of the study and participation requirements, and will be asked to complete an online informed consent (see Human Subjects). Participants will then complete the pretest measures (see Table 3). Upon pretest completion, parents will be randomly assigned to either the APT intervention condition or a content comparison (CC) group.

Content Comparison (CC). Parents assigned to the CC will be given access to a self-paced online training program covering the same content as APT. The CC group will receive an online program that delivers antecedent-behavior-consequence (ABC) multimedia instruction that is targeted to parents. For this purpose, investigators and the curriculum designer will adapt a program developed by IRIS entitled Teaching Routines to Children Who Have ASD, A Parent's Guide to the ABC Method. The ABC Method demonstrated in a pre-posttest design that web-based instruction in applied behavioral analytical (ABA) strategies, such as ABC, was effective in helping parents teach children basic self-help skills, and allowed parents to apply this method to a range of skills. The original ABC Method program consisted of nine multimedia lessons (modeling videos, animated sequences, interactive exercises, downloadable summaries) designed to help parents understand and use the antecedent-behavior-consequence concept derived from ABA. Each lesson contained a 3 to 5 minute video that uses simple language, realistic live action, and animation to illustrate a concept and to model how parents can apply the concept as they teach a routine. Each lesson also contained an interactive exercise and printed summary to guide parents through the steps of creating a teaching plan tailored to the needs of their children.

To ensure that the CC group receives a dosage equivalent to that of the APT Intervention group, the original program will be reformatted so that it is delivered in 3 rather than 9 lessons. This will require re-editing the original materials, creating new introductions to the three lessons, and making corresponding changes in how the program is delivered by our online Learning Management System. Investigators will also ensure that the reformatted program possesses equivalent validity with the original program. Investigators and the development team will achieve this by enlisting a small test group of parents in an iterative process of review and refinement as the program is reformatted. Parents in the CC will have 3 weeks in which to access the program. Web metrics will allow investigators to track adherence to program fidelity.

Treatment. Parents in the APT group will be presented with the dates and times of available training groups and asked to select their preference. They will then receive an access code for logging on to the APT web hub to view the training materials. Participants will also be given access to the videoconferencing workshops, and will test to ensure they can access the site and that their camera and microphone are operating. IRIS Ed technical staff will be available to assist with any difficulties. Each week, for three weeks participants in the APT condition will meet with their training group and the APT Parent Educator for 120 minutes of instruction, discussion, and problem solving. They will also complete assigned homework, including watching online video trainings.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 3-8 who have autism

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nell Caraway, BA, Principal Investigator — IRIS Educational Media; Meme Hieneman, Ph.D., BCBA, Principal Investigator — IRIS Educational Media
Locations (1):
- IRIS Educational Media, Eugene, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Autism Parent Trainer (APT): Autism Parent Trainer (APT) Experimental Condition.
  Practiced Routines was a facilitated program. It was organized into four modules that included a total of seven videos ranging from 3-13 minutes each. The topics overlapped with those in the TR program, but included more explicit information on function-based strategies, as well as mindfulness practice. Participants were assigned six fillable forms, and provided supplemental data collection tools. Additional resources focused on mindfulness and PBS within family routines. Eighteen brief guided audio meditations were available to participants via the Practiced MindTM mobile application. The meditations focused on bringing the parents' awareness to both internal and external experiences and helping them act intentionally.
- Teaching Routines (Control): Teaching Routines was entirely self-directed. The program included eight modules with videos for each ranging 3 - 5 minutes in duration. The topics were antecedent-behavior-consequence method, creating task analyses, antecedent-based strategies, communication, reinforcement, teaching methods, and overcoming obstacles. Participants were assigned six activities using fillable forms and provided additional resources including examples, a glossary of terms, and a list of websites. No feedback was given to the parents apart from the automated completion responses. The participants were given access to the TR LMS for the duration of the study, but post and follow-up assessments were completed at 6 and 10 weeks (i.e., same as the PR condition).
Period: Overall Study
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Started | 77 | 79
Completed | 73 | 72
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control) | Total
Number analyzed (Participants) | 77 | 79 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 79 | 156
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (5.9) | 36.1 (5.5) | 36.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 77 | 152
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 67 | 62 | 129
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 5 | 18
  White | 56 | 66 | 122
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 77 | 79 | 156

OUTCOME MEASURES:

1. Primary Outcome: Child Behavior Measured by Strengths and Difficulties Questionnaire (Goodman, 1997)
Description: Examining change over time points (T2-T1) This 25-item parent-report version of a behavioral screening questionnaire has been used with children aged 3 to 16 years of age. It assesses both positive and negative behaviors in the following domains: conduct problems, inattention-hyperactivity, emotional symptoms, peer problems, and pro-social behavior. The SDQ-P has demonstrated acceptable psychometric properties and is available in Spanish (Goodman, 2001).Total range of scores is from 0 to 50. The prosocial items are reverse scored for the total scale so that on the total scale higher scores indicate worse behaviors.
Time Frame: Pre (0 weeks), Post (3 weeks)
Measure: Mean (Standard Deviation); unit: total score on a scale
Groups:
- Autism Parent Trainer (APT): Autism Parent Trainer (APT) Experimental Condition. This group will receive Google Hangouts training on autism and lifestyle coaching.
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Number analyzed (Participants) | 77 | 79
total score on a scale | 19.27 (5.2) | 21.00 (5.2)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control); To address hypotheses predicting differential change in outcome measures between condition over time we used analysis of covariance (ANCOVA) models that allow for examination of cross-sectional effects and mean adjusted outcomes. The ANCOVA models (adjusted for baseline scores) were used for analyses of change in the outcome measures at posttest; Test type: Superiority; p = .598, ANCOVA

2. Primary Outcome: Family Quality of Life as Measured by Family Quality of Life Survey (Summers et al., 2005)
Description: Examining change over time points (T2-T1) Quality of Life was measured using the Family Quality of Life survey (FQOL; Summers et al., 2005), which is a 25-item measure of the quality of life for a family raising a child with intellectual or developmental disabilities. The outcomes measured are: quality of life in the domains of parenting, emotional well-being, physical/material well-being, and disability-related supports using a 5-point scale with responses ranging from (1) very dissatisfied to (5) very satisfied. The average score on the total scale was used in the analysis. The range is from 1 to 5 with higher scores indicating more positive outcomes.
Time Frame: Pre (0 weeks), Post (3 weeks)
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control
Number analyzed (Participants) | 77 | 79
average score on a scale | 3.99 (.5) | 3.86 (.6)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control; . To address hypotheses predicting differential change in outcome measures between condition over time we used analysis of covariance (ANCOVA) models that allow for examination of cross-sectional effects and mean adjusted outcomes. The ANCOVA models (adjusted for baseline scores) were used for analyses of change in the outcome measures at posttest; Test type: Superiority; p = .81, ANCOVA

3. Primary Outcome: Parenting Scale (Arnold, O'Leary, Wolff, & Aker, 1993)
Description: Examining change over time points (T2-T1) Parenting Practices will be assessed using the Parenting Scale (PS; Arnold, O'Leary, Wolff, & Aker, 1993) a 30-item, 7 point Likert-like scale with three subscales (laxness, over-reactivity, and hostility). The scale has internal consistency for the total scale and subscales (α = .78 and - .83 respectively) and has been evaluated for factor structure and validity (Rhoades & O'Leary, 2007). The average score on the total scale was used in the analysis with a range of 1 to 7 with lower scores indicating more positive outcomes.
Time Frame: Pre (0 weeks), Post (3 weeks),
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Number analyzed (Participants) | 77 | 79
average score on a scale | 3.7 (.6) | 3.72 (.3)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .404, ANCOVA

4. Primary Outcome: Scales of Independent Behavior-Revised (SIB-R; Bruininks, Woodcock, Weatherman, & Hill, 1996)
Description: Examining change over time points (T2-T1)
  The SBI-R is a 40-item, 7-point scale that measures 14 areas of adaptive behaviors and 8 areas of maladaptive behaviors.
  We used the total adaptive scale with a total range of 0 to 120 with higher scores indicating better outcomes.
Time Frame: Pre (0 weeks), Post (3 weeks)
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Number analyzed (Participants) | 77 | 79
total score on a scale | 65.56 (15.4) | 63.87 (16.2)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .246, ANCOVA

5. Secondary Outcome: Knowledge About Applied Behavior Analysis and Acceptance Commitment Training Measured by Questionnaire
Description: Examining change over time points (T2-T1) 20 multiple choice knowledge items were developed during the project and were used to determine the extent to which participants understood basic program content, e.g., techniques parents can use to help their child master self-care routines. These included questions about the principles of behavior support (gathering information, evaluating possible reinforcers, etc.), definitions of behavioral concepts (tantrums, reinforcement, antecedent), and application of these concepts. The total score ranged from 0 to 20 with higher scores indicating better outcomes.
Time Frame: Pre (0 weeks), Post (3 weeks)
Measure: Mean (Standard Deviation); unit: total correct answers
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Number analyzed (Participants) | 77 | 79
total correct answers | 14.52 (2.7) | 13.37 (2.4)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .007, ANCOVA

6. Secondary Outcome: Consumer Satisfaction Questionnaire
Description: A 16-item scale was developed to evaluate parents' views of the feasibility, usability, and personal relevance of the program. It asked about the information taught in the program, the trainers, the website, and the other materials. The average score on these 19 items was evaluated and ranged from 1 to 6 with higher scores indicating more positive outcomes.
Time Frame: Follow up (6 weeks)
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
Number analyzed (Participants) | 77 | 79
average score on a scale | 5.50 (.67) | 5.24 (.88)
Statistical Analysis 1: Comparison: Autism Parent Trainer (APT) vs Teaching Routines (Control); Two-sample t-test; Test type: Superiority; p = .045, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Six weeks from pretest to follow-up.
Description: This was a self-selected behavioral training program for parents of children with Autism.
Arm/Group | Autism Parent Trainer (APT) | Teaching Routines (Control)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/79
Other Adverse Events (participants affected / at risk) | 0/77 | 0/79

LIMITATIONS AND CAVEATS:
The most significant limitation of this study was that it was underpowered for a content comparison study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT02469870/Prot_SAP_000.pdf